CLINICAL TRIAL: NCT07259135
Title: Hemorrhagic Risk and Hemostasis Disorders in Noonan Syndrome and Related Conditions
Brief Title: Link Between Abnormal Bleeding and Coagulation Disorders in Noonan Syndromes
Acronym: PlatNoon
Status: Not yet recruiting | Type: Observational
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Other Study IDs: CHUBX 2024/96
Record Dates: First submitted 2025-07-22; First posted 2025-12-02 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Noonan Syndrome
Keywords: Noonan; Retrospective; Prediction; Hemorrhagic; Hemostasis; Bleeding; Surgery
MeSH Terms: conditions — Noonan Syndrome; Hemorrhage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Noonan Syndrome (SN): Cohort of SN patients meeting study eligibility criteria
  Interventions: Other: Reuse of routine clinical and biological data

INTERVENTIONS:
Other: Reuse of routine clinical and biological data — Reuse of routine clinical and biological data

SUMMARY:
Noonan syndrome is a relatively rare genetic disorder, affecting around 1 in every 1,000 to 2,500 children born. Patients often have a tendency to bleed more easily, particularly from the skin or mucocutaneous tissue (such as mouth or nose). Around half of all the patients are affected by bleedings. The causes of bleeding are variable : some are linked to platelet disorders, others to more complex coagulation problems. However, it is difficult to predict exactly which patients are at risk of severe bleeding, for example during surgery. This is why there are as yet no clear recommendations for preventing this risk before medical intervention. However, it is recommended that patients with Noonan syndrome consult a specialist to assess this risk. Unfortunately, the tests carried out are often unreliable in predicting this significant risk of bleeding. In this study, data from a large group of patients with Noonan syndrome, followed-up in different centers in France, will be studied. During a medical meeting as part of their regular follow-up, a medical doctor assessed their tendency to bleed using a standardized questionnaire (standardized ISTH-BAT score). These results will be compared with the biological tests also performed during their medical follow-up. The aim is to better understand whether these tests are useful in predicting the risk of bleeding. Ultimately, this could help practicians to better anticipate surgical or medical interventions in these patients, and limit bleeding-related risk.

DETAILED DESCRIPTION:
Noonan syndrome (NS) is an autosomal dominant genetic disorder, with an estimated prevalence of 1 in 1,000 to 2,500 births/year. Patients with NS have a cutaneous-mucosal hemorrhagic diathesis, with a prevalence estimated at 46% in a large meta-analysis. The most frequently reported abnormalities are those of primary hemostasis (thrombocytopenia, thrombopathy and Willebrand's disease), as well as those of coagulation, but the correlation between symptomatology and hemostatic disorders is unclear. As a result, there are no specific recommendations in terms of intraoperative hemorrhagic risk prevention, due to a lack of knowledge of the real hemorrhagic risk in these patients, who are particularly exposed to invasive procedures. The PNDS recommends that patients be referred to a haemostasis specialist for assessment of bleeding risk, which entails the performance of investigations that are often not very predictive of bleeding risk. Interpretation of these results with regard to bleeding risk therefore remains unsolved. It is against this backdrop that the aim of this study is to retrospectively collect the bleeding diathesis of a national cohort of patients with SN, using a standardized ISTH-BAT score, performed in the context of a specialized hemostasis consultation by a physician from one of the centers involved in this study. The hemorrhagic diathesis will be compared with the results of the hemostasis exploration performed as part of their follow-up (routine care). This study will make it possible to assess the value of a hemostasis study in predicting the risk of bleeding in these patients.

ELIGIBILITY:
Inclusion Criteria:

* All patients with SN, regardless of age
* Patient/parental guardians informed of the study
* Patient/legal representative not opposed to the use of their/the child's data
* Person affiliated or benefiting from a social security scheme

Exclusion Criteria:

- Adults protected by law (guardianship, curatorship or safeguard of justice)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patient with noonan syndrome
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2027-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
ISTH-BAT haemorrhagic score | At first clinical visit in the referent center (retrieved retrospectively at inclusion visit)
  The ISTH-BAT standardized questionnaire uses 14 items to assess the severity of cutaneous-mucosal, cerebral, articular and per- or post-operative haemorrhagic symptoms
Willebrand factor | At first clinical visit in the referent center (retrieved retrospectively at inclusion visit)
  The Willebrand factor will be obtained from biological tests (in percentage of controls mean value)
Platelet function | At first clinical visit in the referent center (retrieved retrospectively at inclusion visit)
  Platelet function will be obtained from biological tests (in percentage of controls mean value)

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Bordeaux, Service Hématologie Biologique, Bordeaux, France

IPD SHARING:
Plan to Share IPD: No